CLINICAL TRIAL: NCT01904331
Title: Study of the Cardiovascular and Psychosocial Effects of the Treatment of Breast Cancer With Chemotherapy and/or Radiotherapy
Brief Title: Breast Cancer Long-term Outcome of Cardiac Dysfunction
Acronym: BLOC
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dr. A.J. Berendsen, Dr., University Medical Center Groningen
Other Study IDs: 686317
Record Dates: First submitted 2013-07-11; First posted 2013-07-22 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Breast Neoplasms
Keywords: Cardiotoxicity; long-term effects; chemotherapy; radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — EDTA-plasma, Heparin-Lithium plasma, Serum, Frozen whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer patients: Women who were curatively treated with chemo- and/or radiotherapy for breast cancer
- Controls: Women matched on age and general practitioner with the breast cancer patients

SUMMARY:
The purpose of this study is to assess the prevalence of cardiac dysfunction and (undiagnosed) heart failure in women registered in general practice with a history of breast cancer who received chemotherapy and / or radiotherapy as compared to a matched female control population.

DETAILED DESCRIPTION:
Background:

Due to screening and progress in treatment the overall survival of women treated for breast cancer has increased over the last decades. Therefore, the long-term effects of breast cancer have emerged as an important topic. An increased mortality is seen within years post treatment due to an increased incidence of cardiac dysfunction among survivors of breast cancer. This increased mortality is related to long term side effects of treatment with chemotherapy and radiotherapy. Earlier studies into this topic have focused on specific patient groups and therefore these results are difficult to translate to the general population. Furthermore, most echo graphic studies have focused on the systolic dysfunction of the heart, which is a late stage of the cardiac deterioration. Detecting cardiotoxicity early on provides the opportunity for early treatment and might therewith prevent deterioration of cardiac function and improve the prognosis of patients

Objectives:

Primary objective

1. To assess the risk of a systolic and / or diastolic cardiac dysfunction at echocardiography of breast cancer patients compared to matched controls.

   Secondary objective:
2. To assess the risk of heart failure( a combination of clinical complaints, objective measures at physical examination, laboratory examination or echocardiography) in breast cancer patients as compared to matched controls
3. To determine the value of patient characteristics, clinical complaints and signs in physical examination in diagnosing cardiac dysfunction as found of echocardiography
4. To determine the additional diagnostic value of biomarkers; N-terminal pro-hormone of brain natriuretic peptide (NT-pro-BNP) and high sensitive troponin T (hs-troponinT) in diagnosing cardiac dysfunction, as found on echocardiography
5. Genetic analysis

Study design and population:

This is a cross-sectional, observational study in women in general practice who have been curatively treated for breast cancer with chemo and / or radiotherapy at a minimum of 5 years ago and an age and general practitioner (GP) matched female control population. Patients must be 18 years or older, younger than 80 at the time of diagnosis, not been treated for other types of cancer with chemo- and/or radiotherapy and must be willing to give written informed consent Primary study parameters

1. Systolic and diastolic cardiac function of echocardiography
2. Hospital Anxiety and Depression Scale (HADS)
3. Multi dimensional Fatigue Inventory (MFI-20)
4. Cardiovascular Risk Management (CVRM)
5. Short physical examination: blood pressure, height, weight, waist circumference, electrocardiography, signs of edema, auscultation
6. Laboratory testing: Hemoglobin, hematocrit, leucocytes, creatinine , estimated glomerular filtration rate (GFR), cholesterol, triglycerides, High-density lipoprotein (HDL) cholesterol, Low-density lipoprotein (LDL) cholesterol, Cholesterol/HDL ratio, C-reactive protein (CRP),Thyroid stimulating hormone (TSH), glucose
7. Serum and plasma for biomarkers
8. ethylenediaminetetraacetic acid (EDTA) -tube for DeoxyriboNucleic Acid (DNA) analysis Outcomes

Primary outcome:

The cardiac dysfunction will be related to type of therapy and compared to the age-and general practice matched control group. Information on type of therapy will be gathered trough contacting the hospitals were patients were treated.

Secondary outcome:

Symptoms and signs of women with cardiac dysfunction will be compared with those without cardiac dysfunction. A comparison between women treated for breast cancer and women without breast cancer will be made.

The level of the biomarkers will be linked with the cardiac dysfunction. In women treated for breast cancer with chemo- and/or radiotherapy these will also be linked with type of therapy.

DNA analysis will be carried out to investigate if changes in candidate genes are related to the development of cardiac dysfunction.

Burden and risks associated with participation, benefit and group relatedness The minimal invasive tests will be performed if patient are willing to participate in de study after contact trough letters. As far as known no serious adverse events are linked to the described study procedures.

With this study we hope to get insight in the risk of cardiac dysfunction after chemo- and/or radiotherapy in women treated for breast cancer. And to determine possibly diagnostic measure to detect this deterioration. Eventually, this may contribute to the early detection of cardiac dysfunction in women treated with chemo- and/or radiotherapy for breast cancer to improve the prognosis for patients.

ELIGIBILITY:
Inclusion Criteria:

* For breast cancer patients: minimum of 5 years after treatment for breast cancer with chemo- and/or radiotherapy and after 1970
* For breast cancer patients: younger than 80 at the time of diagnosis of breast cancer
* willing to sign an informed consent
* older than 18 at the time of inclusion

Exclusion Criteria:

* Treatment with chemo- and/or radiotherapy for other types of cancer besides breast cancer
* women who are unable to participate (e.g. terminally or mentally ill)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients are selected in primary care practices in the Northern part of the Netherlands.
  Controls are randomly selected in the same primary care clinics as participants.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02-06 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Cardiac dysfunction | on average 11 years after treatment with breast cancer
  systolic and diastolic parameters at time of inclusion

SECONDARY OUTCOMES:
Biomarkers +DNA | on average 11 years after treatment with breast cancer
  Plasma EDTA, lithium-heparin plasma and serum are stored at -80 freezer at the the time of inclusion. Determination of biomarkers will take place at the end of the study period Whole blood is frozen for DNA analysis at time of inclusion.

OTHER OUTCOMES:
Clinical complaints and signs at inclusion | on average 11 years after treatment with breast cancer
  Questionnaires (CVRM, HADS and MFI-20), a short physical examination and a electrocardiography at time of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Y Berger, M.D. Ph.D., Study Director — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen (UMCG), Groningen, Netherlands